CLINICAL TRIAL: NCT03326908
Title: Description of the Interdigitation Retinal Area by SD-OCT (Spectral Domain Optical Coherence Tomography): An Exploratory Study (ODIGIT)
Brief Title: Description of the Interdigitation Retinal Area by SD-OCT: An Exploratory Study
Acronym: ODIGIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MMT_2017_16
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2018-01

CONDITIONS: Tomography, Optical Coherence; Retina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal conditions of light exposure (Other): Spectral Domain Optical Coherence Tomography (SD-OCT):
  Five SD-OCTs will be produced under the same lighting conditions (photopic).
  * At baseline
  * 20 minutes after baseline
  * 25 minutes after baseline
  * 45 minutes after baseline
  * 60 minutes after baseline
  Interventions: Device: Spectral Domain Optical Coherence Tomography
- Light variations (Other): Spectral Domain Optical Coherence Tomography (SD-OCT):
  Five SD-OCT will be performed:
  * at baseline, in a room with photopic artificial lighting (400 lux)
  * after a period of adaptation to the dark (20 minutes in the dark: 0 lux)
  * after 5 min of retinal glare, obtained by means of a projection of light of 1000 lux on the fundus of eye
  * 15 minutes after this period of retinal glare, in photopic artificial lighting
  * 30 minutes after the period of retinal glare, in photopic artificial lighting
  Interventions: Device: Spectral Domain Optical Coherence Tomography

INTERVENTIONS:
Device: Spectral Domain Optical Coherence Tomography — Five SD-OCTs will be performed with various conditions of enlightenment.

SUMMARY:
Improvement of retinal medical imaging opens new perspectives for exploring the retinal structures. Optical coherence spectral domain (SD-OCT), which has been widely used in the last ten years, is certainly the most advanced device. In the analysis of patients without retinal disease using SD-OCT, granulations in the interdigitation area were observed. These granulations have never been described with this device. They could correspond either to the degradation products of the external segments of the photoreceptors or to melanosomes. A descriptive study of these granulations at different examination times and in different lighting situations would allow us to obtain essential information for a better understanding of this area. Based on the results, larger studies could explore this area more finely in retinal pathologies involving dysfunctions of photoreceptors or of the pigmentary epithelium.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Consent to participate

Exclusion Criteria:

* Retinal abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Variation of the number of hyperreflective granulations in the interdigitation area according to time and enlightenment | 1 hour after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathis T, Vasseur V, Zuber K, Arej N, Loria O, Kodjikian L, Sennlaub F, Mauget-Faysse M. Light-induced modifications of the outer retinal hyperreflective layers on spectral-domain optical coherence tomography in humans: an experimental study. Acta Ophthalmol. 2021 Nov;99(7):765-772. doi: 10.1111/aos.14723. Epub 2021 Jan 4. PMID 33393736